CLINICAL TRIAL: NCT06719895
Title: Web-Based Newborn Care Education for Primiparous Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Veysel Can, Asst. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: web based
Record Dates: First submitted 2024-11-19; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Web Based Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web based education (Experimental)
  Interventions: Behavioral: web based education
- control (No Intervention)

INTERVENTIONS:
Behavioral: web based education — experimental
  Arms: web based education

SUMMARY:
For pregnant women expecting their first baby, readiness during pregnancy is an important factor in successfully performing hygienic care for their babies. This study was planned to determine the effect of web-based education on the readiness levels of primiparous pregnant women for newborn hygienic care practices. In this study, the aim was to support pregnant women and mothers after birth in newborn care and to develop their application skills with the web-based education program given to primiparous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 15 and 19 years
* Being 19 years old and above
* Being literate
* Being primigravida
* Having a single baby (not twins or more)
* Being a volunteer to participate in the study
* Having no health problems for the mother and the baby
* Having a computer, tablet or smart phone and the ability to use it
* Having regular internet access

Exclusion Criteria:

* The mother being 18 years of age or younger
* Being multigravida and/or multiparous
* Having a health problem related to the mother or the baby
* Not having a smart phone or wireless internet during the study period
* Not filling out the survey forms incompletely and not watching videos about hygienic care of the newborn

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Mothers' readiness levels for hygienic care of newborns | first test and final test 4 weeks after the first test, one month
  Mothers' readiness levels for hygienic care of newborns

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)